CLINICAL TRIAL: NCT00004844
Title: Randomized Study of Fetal Neurotransplantation for the Treatment of Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: University of Colorado, Denver (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13940; UCHSC-COMIRB-9397
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Parkinson Disease; Neurologic Manifestations; Mental Disorders; Rare Diseases

INTERVENTIONS:
Procedure: tissue implantation

SUMMARY:
OBJECTIVES:

I. Assess the safety and efficacy of embryonic mesencephalic dopamine cell implants into the putamen of patients with Parkinson's disease.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind, placebo controlled study. Patients are stratified by age (over and under 60). Patients are randomized to receive either sham surgery or tissue implantation.

Embryonic tissue is prepared. While patients are awake, but sedated, bilateral incisions are made in the skin and burr holes drilled in the skull. A cannula is inserted into the brain to the posterior putamen. Implant patients receive embryonic neural tissue or sham patients have no needles penetrate the brain. After 1 year, patients who receive the sham operation in the first operation may receive embryonic neural tissue in a second operation.

Patients are followed every 4 months during the first year and every 6 months thereafter.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Idiopathic Parkinson's disease for at least 7 years with rest tremor or bradykinesia and one of the following cardinal signs: Rigidity Flexed posture Loss of postural reflexes Freezing (motor blocks)
* Continuing response to levodopa
* Presence of at least one of the following intractable symptoms or signs: Intractable disabling fluctuations Intractable disabling dyskinesias Intractable "on" freezing (i.e., motor blocks that interfere with walking despite being "on"
* Bilateral parkinsonism when "off" (may be asymmetry between right and left sides)
* Decreased dopa uptake in the striatum

--Prior/Concurrent Therapy--

* No prior brain surgery

--Patient Characteristics--

* Cardiovascular: No severe cardiopulmonary disease
* Neurologic: No history of strokes No neuroleptics No encephalitis No oculogyric crisis No remission No cerebellar signs No dementia (Mini-Mental state score no greater than 22) No supranuclear gaze palsy No Babinski sign No orthostatic hypotension No hydrocephalus No brain tumor No occlusive cerebrovascular disease
* Pulmonary: Absolute standing pressure at least 90/60 mmHg
* Other: No diabetes mellitus No exposure to toxins No other severe medical disease Hamilton Depression Scale score of less than 20 points

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 1998-07

CONTACTS AND LOCATIONS:
Overall Officials: Curt R. Freed, Study Chair — University of Colorado, Denver